CLINICAL TRIAL: NCT02198560
Title: RS-3000 Lite Agreement Study
Status: Completed | Type: Observational
Sponsor: Nidek Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: NRL-1
Record Dates: First submitted 2014-07-17; First posted 2014-07-23 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
Keywords: Normal (Eyes without pathologies)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normal (Eyes without pathology)
  Interventions: Device: RS-3000 Lite

INTERVENTIONS:
Device: RS-3000 Lite

SUMMARY:
The primary objectives of the study are to assess the agreement between the two different scan mode of the RS-3000 Lite.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who do not have pathology in both eyes

Exclusion Criteria:

Subjects who have any of the following conditions:

* Diabetes mellitus (DM) and/or diabetic retinopathy
* Uncontrolled Hypertension (HT)
* Cerebral infarction, cerebral hemorrhage, cranial nerve neoplasm and other central nervous system diseases affecting vision
* Cardiac, hepatic, renal and hematologic diseases
* A current condition requiring systemic administration of steroid
* A history of, or currently receiving, anticancer therapy
* Epileptic seizures which are optically induced
* Dementia

Note: Additional criteria may apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal (Eyes without pathology)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-08; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Retinal thickness and Optic Disc Analysis | 3 hours
  Time frame is the maximum duration of hospital stay.

SECONDARY OUTCOMES:
Number of participants with adverse events | 1day

CONTACTS AND LOCATIONS:
Locations (1):
- Nabeta Ganaka Iin, Okazaki, Aichi-ken, Japan